CLINICAL TRIAL: NCT00003659
Title: A Phase II Study of Fludarabine Induction With Sequential High Dose Cyclophosphamide and Rituximab as Consolidation Therapy for Previously Untreated Patients With Intermediate and High-Risk Chronic Lymphocytic Leukemia
Brief Title: Fludarabine, Cyclophosphamide, and Rituximab in Treating Patients Who Have Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 98-080; MSKCC-98080; NCI-G98-1483
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2012-12-31 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-09

CONDITIONS: Leukemia
Keywords: stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Filgrastim; Rituximab; Cyclophosphamide; fludarabine phosphate

ARMS (1):
- intermediate or high risk chronic lymphocytic leukemia (Experimental): This is a single-arm open-label pilot study designed to assess the antileukemic activity of a regimen containing sequential administration of fludarabine, high-dose cyclophosphamide, and rituximab.
  Interventions: Biological: filgrastim; Biological: rituximab; Drug: cyclophosphamide; Drug: fludarabine phosphate

INTERVENTIONS:
Biological: filgrastim — Filgrastim (300 μg for patients ≤ 70 kg or 480 μg for patients > 70 kg) will be administered beginning two days after each cyclophosphamide dose and given for a total of eight subcutaneous daily doses.
Biological: rituximab — Approximately four weeks after the completion of the last cyclophosphamide dose, patients will receive rituximab 375mg/m2 as an intravenous infusion once weekly for four doses.
Drug: cyclophosphamide — Cyclophosphamide 3000mg/m2 will be given intravenously q 2 - 3 weeks x 3 doses.
Drug: fludarabine phosphate — Fludarabine will be administered intravenously at a dose of 25 mg/m2 per day x 5 days every 4 weeks.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells. Monoclonal antibodies can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells.

PURPOSE: Phase II trial to study the effectiveness of fludarabine plus high-dose cyclophosphamide and rituximab in treating patients who have previously untreated chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate in patients with chronic lymphocytic leukemia treated with sequential fludarabine, high dose cyclophosphamide, and rituximab.
* Survival up to 5 years
* Utilize flow cytometry and polymerase chain reaction as sensitive measures of minimal residual disease in these patients.

OUTLINE: This is an open label study.

Patients receive fludarabine IV once daily for 5 days. Treatment is repeated every 4 weeks for 3 or 6 courses.

Three weeks later, cyclophosphamide is administered intravenously every 2-3 weeks for 3 courses. Filgrastim (G-CSF) is administered on days 2-10. Beginning 4 weeks after the last dose of cyclophosphamide, patients receive rituximab by intravenous infusion once weekly for 4 weeks.

Patient are followed every 3 months until death.

PROJECTED ACCRUAL: This study will accrue 30 patients within 3 years.

ELIGIBILITY:
Inclusion criteria:

* Patients must have either intermediate or high-risk chronic lymphocytic leukemia as defined by the three-stage Rai system (see section 2.2 page 2). Patients with Rai intermediate risk disease should meet the criteria for active disease as outlined by the NCI Working Group guidelines (including weight loss, fatigue, fevers, evidence of progressive marrow failure, splenomegaly, progressive lymphadenopathy, or progressive lymphocytosis with a rapid doubling time).
* Patients must be previously untreated (with cytoreductive agents) for their CLL.
* The patient must have an absolute lymphocytosis in the blood of at least 5,000 lymphocytes/μl, or bone marrow lymphocytosis greater than or equal to 30% of all nucleated cells. These lymphocytes must have an appropriate immunophenotype for CLL including expression of CD5 and CD20.
* Karnofsky performance status equal to or greater than 60% (see Appendix B).
* Eligible patients should have a reasonable life-expectancy greater than four weeks.
* Age ≥ 18 years and ≤ 75 years.
* Total bilirubin ≤ 2.0 mg per deciliter. Total creatinine ≤ 2.0 mg/ dl.
* Platelet count ≥ 50,000/ ul.
* Signed informed consent, which indicates the investigational nature of this, is required.
* No patient may be entered onto the study without consultation with the principal investigator.

EXCLUSION CRITERIA:

* Patients with Rai intermediate risk disease who meet the criteria of Montserrat "smouldering leukemia" will not be eligible for treatment on this protocol.
* Patients with significant autoimmune hemolytic anemia or autoimmune thrombocytopenia shall not be eligible for treatment on this protocol as there is some evidence that fludarabine can worsen these conditions.
* Patients with active infections requiring systemic antibiotics.
* Prior cytotoxic treatment of their CLL.
* Pregnant or lactating women. Women and men of childbearing age should use effective contraception.
* Patients with a serious cardiac condition.
* Concomitant chemotherapy or radiotherapy while on protocol.
* Concomitant prednisone therapy will not be permitted as the combination of fludarabine and prednisone is known to increase the risk of opportunistic infections. Patients may receive intravenous immunoglobulin (IVIG) and other supportive care measures as clinically appropriate while on protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 1998-09; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Adam Weiss, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual 09/08/1998 Protocol Closed to Accrual 06/14/2005 Primary Completion Date 05/12/2009 Recruitment Location is the medical clinic
Period: Overall Study
Arm/Group | Intermediate or High Risk Chronic Lymphocytic Leukemia
Started | 39
Completed | 36
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Intermediate or High Risk Chronic Lymphocytic Leukemia
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 31
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Response was determined as indicated in the protocol. The categories are: complete response, nodular partial response, partial response and failure. The major criteria for determination of response to therapy in patients with CLL include physical examination and examination of the peripheral blood and bone marrow. The laboratory and radiographic studies which were abnormal pre-study, will be repeated to document the degree of maximal response.
Time Frame: 3 years
Population: There were 36 assessable patients as described in the protocol
Measure: Number; unit: participants
Arm/Group | Intermediate or High Risk Chronic Lymphocytic Leukemia
Number analyzed (Participants) | 36
participants
  Complete Response | 22
  Nodular Partial Response | 2
  Partial Response | 8
  Failure | 4

2. Secondary Outcome: Utilize Flow Cytometry and Polymerase Chain Reaction as Sensitive Measures of Minimal Residual Disease
Description: The flow cytometric response and the molecular polymerase chain reaction (PCR) response was captured as indicated in the protocol. Immunophenotypic analysis of bone marrow and/ or peripheral blood demonstrate a normal k:λ ratio and a normal number of CD5/CD19 (or CD5/CD20) dual staining cells (<5% of the lymphocyte gate).
Time Frame: 3 years
Population: All assessable patients as indicated in the protocol
Measure: Number; unit: participants
Arm/Group | Intermediate or High Risk Chronic Lymphocytic Leukemia
Number analyzed (Participants) | 36
participants
  Flow cytometric complete response | 20
  Molencular (PCR) complete response | 12

3. Secondary Outcome: Overall Survival Status
Description: The 5 year survival rate. The survival of patients with this disease is dependent on the stage of disease. Two useful staging systems are: Three-stage Rai System Clinical Feature and the Binet System.
Time Frame: up to 5 years
Population: All assessable patients as indicated in the protocol.
Measure: Number; unit: participants
Arm/Group | Intermediate or High Risk Chronic Lymphocytic Leukemia
Number analyzed (Participants) | 36
participants | 26

ADVERSE EVENTS:
Arm/Group | Intermediate or High Risk Chronic Lymphocytic Leukemia
Serious Adverse Events (participants affected / at risk) | 10/36
Other Adverse Events (participants affected / at risk) | 32/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intermediate or High Risk Chronic Lymphocytic Leukemia (N=36)
Anemia (Blood and lymphatic system disorders) | 6
Pulmonary, other Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2
Infection with grade 3/4 neut (Infections and infestations) | 5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intermediate or High Risk Chronic Lymphocytic Leukemia (N=36)
Neutropenia (Blood and lymphatic system disorders) | 32
Thrombocytopenia (Blood and lymphatic system disorders) | 28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes